CLINICAL TRIAL: NCT05353023
Title: Intensive Care Unit Activity in France From the National Database Between 2013 and 2019: More Critically Ill Patients, Shorter Stay and Lower Mortality Rate
Brief Title: Intensive Care Unit Activity in France From the National Database Between 2013 and 2019
Acronym: ICU_ACTIVITY
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2022/JYL-01
Record Dates: First submitted 2022-04-25; First posted 2022-04-29 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2022-04

CONDITIONS: Critical Illness; Intensive Care Unit
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ICU ADMISSION: All patients admitted in a French intensive care unit over a 7-year period (2013 to 2019) using the French National Uniform Hospital Discharge Database (PMSI)

SUMMARY:
Using data from the French National Uniform Hospital Discharge Database (systematically collecting administrative and medical information related to all hospitalized patients in France for care reimbursement purposes), the present study retrospectively assesses the activity of the French Intensive Care Unit (ICU)(1,594,801 ICU admissions):

* In-ICU and in-hospital mortality rates
* Length of stay in ICU and hospital
* Mortality-associated factors during the study period.
* Number of organ failures
* Bed occupancy,
* Regional variations in previous indicators

ELIGIBILITY:
Inclusion Criteria:

All adults patients admitted in French ICU between January 1st, 2013, to December 31st, 2019

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adults patients admitted in French ICU between January 1st, 2013, to December 31st, 2019
Sampling Method: Non-Probability Sample
Enrollment: 1594801 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Evolution in mortality rate | from January 1st, 2013, to December 31st, 2019
  evolution of the mortality rate of ICU patients over the study period (2013-19)
Evolution in organ failure rate | from January 1st, 2013, to December 31st, 2019
  evolution of the organ failure rate of ICU patients over the study period (2013-19)
Evolution in ICU stay | from January 1st, 2013, to December 31st, 2019
  evolution of the ICU stay of ICU patients over the study period (2013-19)
Evolution in SAPS (Simplified Acute Physiology Score) II score at admission | from January 1st, 2013, to December 31st, 2019
  evolution of the SAPS II score at admission of ICU patients over the study period (2013-19)
Evolution in age at admission | from January 1st, 2013, to December 31st, 2019
  evolution of the age at admission of ICU patients over the study period (2013-19)
Evolution in sex ratio | from January 1st, 2013, to December 31st, 2019
  evolution of the sex ratio of ICU patients over the study period (2013-19)

SECONDARY OUTCOMES:
Proportion of patients admitted in ICU with at least 2 different organ failures | from January 1st, 2013, to December 31st, 2019
  evolution of the proportion of patients admitted in ICU with at least 2 different organ failures corresponding to the definition of ICU in France.
- Proportion of patients admitted in ICU with a SAPS II score over 15 and with a specific ICU supportive therapy | from January 1st, 2013, to December 31st, 2019
  Evolution of the proportion of patients admitted in ICU with a SAPS II score over 15 and with a specific ICU supportive therapy leading to a reimbursement by the French national health insurance.
Factors Associated with in-ICU mortality | from January 1st, 2013, to December 31st, 2019
  Effect of year-time on in-ICU mortality
Regional variations | from January 1st, 2013, to December 31st, 2019
  Evolution and potential differences between French regions in admission level

CONTACTS AND LOCATIONS:
Overall Officials: Jean Yves LEFRANT, Principal Investigator — Centre Hospitalier Universitaire de Nīmes
Locations (1):
- Intensive care Unit CHU Nîmes, Nîmes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Boulet N, Boussere A, Mezzarobba M, Sofonea MT, Payen D, Lipman J, Laupland KB, Rello J, Lefrant JY, Muller L, Roger C, Pirracchio R, Mura T, Boudemaghe T. Intensive Care Unit activity in France from the national database between 2013 and 2019: More critically ill patients, shorter stay and lower mortality rate. Anaesth Crit Care Pain Med. 2023 Oct;42(5):101228. doi: 10.1016/j.accpm.2023.101228. Epub 2023 Apr 7. PMID 37031815